CLINICAL TRIAL: NCT05057260
Title: LOng COvid Multidisciplinary Consortium: Optimising Treatments and servIces Across the NHS (LOCOMOTION)
Acronym: LOCOMOTION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Collaborators: Imperial College London (Other); University of Oxford (Other); University of Exeter (Other); King's College London (Other); University of Manchester (Other); University of Dundee (Other); Leeds Comunity Healthcare NHS Trust (Other); Oxford University Hospitals NHS Trust (Other); Imperial College Healthcare NHS Trust (Other); University Hospitals, Leicester (Other); Birmingham Community Healthcare NHS (Other Government); NHS Tayside (Other Government); Newcastle-upon-Tyne Hospitals NHS Trust (Other); University Hospital of Wales (Other)
Responsible Party: Principal Investigator, Dr Manoj Sivan, Associate Professor and Consultant in Rehabilitation Medicine, University of Leeds
Other Study IDs: 303623
Record Dates: First submitted 2021-09-23; First posted 2021-09-27 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long Covid cohort: Long Covid patients managed in the 10 participating sites
  Interventions: Other: No drug invervention

INTERVENTIONS:
Other: No drug invervention — No clinical trial

SUMMARY:
Background: Long Covid (LC) affects over one million people in the UK, it has various symptoms and impacts daily life. Although there are 83 LC clinics in England, most people have not had access to them, and waiting times to be seen are long. We realise the urgency for LC patients to access prompt and appropriate care in clinics and doctors' surgeries, as well as manage their symptoms effectively at home.

Aim:Our research aims to produce a 'gold standard' for care by analysing what is happening to patients now, creating new systems of care and evaluating them to establish best practice.

Outline Of Research: This research has been developed with LC patients and will continue to include patients working as equal partners. Key priorities of LC patients are: correct clinical assessment; advice and treatment; and help with returning to work and other roles. This research is also based on the experience of a wide range of NHS professionals already treating people in ten LC clinics across the UK, and led by academics (universities) with links to other LC funded studies.

The research will take place in three settings: LC clinics; at home (including self-monitoring on a mobile device using a set of questions on symptoms built into an app); and in doctors' surgeries. We will track where patients are being referred or not referred, and learn from the experience of clinics by interviewing patients and recording outcomes. Throughout, specialists in 'Healthcare Inequality' will reach people who are not accessing clinics. We will put in place new processes in clinics and doctors' surgeries, monitored throughout to make sure they are the correct standard, accessible for patients and staff, and cost-effective.

Outcomes: Comparing findings across our partnership of ten LC Clinics we will learn more about treatment, providing real-time education to other healthcare staff and patients, and establishing a 'gold standard' that can be shared within England and the rest of the UK.

DETAILED DESCRIPTION:
Background: Long COVID (LC) or Post-COVID syndrome affects up to one million people in the UK and is a syndrome of persistent and fluctuating symptoms, with underlying organ dysfunction and multimorbidity. England has 83 dedicated multidisciplinary LC clinics (with no funding yet in Scotland, Wales or Northern Ireland), but these are unable to meet the growing demand and many patients are currently not getting timely care. There is an urgent need to develop a UK-wide efficient integrated LC service.

Aim: We will optimise LC management across three settings of care - LC specialist clinics (Work stream (WS)1); Homes/self-management (WS2) and Primary care (WS3).

Methods: WS1: The management options for multisystem medical problems will be standardised to derive best practice guidance using a Quality Improvement collaborative involving embedded clinician researchers from 10 UK-wide LC clinics. Experience-based co-design with patients and healthcare professionals will inform training and resources for both. Ethnic and socioeconomic inequalities of care and vocational challenges of patients will be addressed using qualitative and mixed methods approaches.

WS2: A digital platform incorporating wearable technology will capture symptom fluctuations and individual condition triggers to enable biofeedback for self-management. Core outcomes measures including the first published LC patient-reported outcome measure (Yorkshire Rehabilitation Scale C19 YRS, developed by the co-CI) will be made available on the digital platform for monitoring and directing interventions remotely.

WS3: Existing primary care and LC clinic integrated data will assist in developing and evaluating new integrated cost-effective service models that will enable the best practice guidance developed in WS1 to be delivered at point of contact in primary care. We have links with previously funded NIHR LC projects to enable co-learning and maximising impact.

PPI/E: From understanding how COVID-19 has disproportionately affected different communities, we have created a seven-member core PPI Advisory Group (PAG) that is inclusive of different cultural, ethnic and socio-economic groups. They have attended our proposal research planning meetings and met separately to examine and develop the research aim/objectives/ questions, ensuring these are aligned with the key research priorities of patients with LC as well as representing different patient needs.

PAG members have lived experience of LC, and bring information and experience from participating in patient support groups including Long Covid Support (n=38K), doctors with LC and a LC Physio. PAG members have been involved in research design for previous NIHR bids, have acted as patient representatives on the NHS England LC Taskforce, and have led national audits on access to LC clinics. The PPI Lead is a founding member of the LC Employment Taskforce of Society of Occupational Medicine and a representative on the Access to WHO Covid Therapies Accelerator (ACT-A) committee. Some members meet weekly as members of Employment Steering Group of the LC Support Group including liaising with Unions.

In this study, the PAG will meet quarterly to review progress, ensure the research is answering the most relevant urgent issues in LC care and that the findings are translational and rapidly informing LC care. To ensure the different demographics of each of the ten LC Clinics are represented, two PPI members from each Clinic will be invited to join a Patient Advisory Network (PAN). Information will flow between the PAG and the PAN via the PPI Lead and Co-lead, ensuring that the voices of the PAN are represented within the PAG, and that they receive updates about research activity in the same way as PAG members. With support from the PPI Lead and Co-lead, PAN members will have an active role in gathering and sharing local intelligence about various aspects of the LC experience and LC Clinic access from LC patients representative of different groups e.g. via the voluntary sector and GP surgeries in different locations, including remote areas where there may be more elderly people with less access to LC clinics. The PPI Facilitator will provide the PAN members with PPI training, and provide them with the appropriate support needed to carry these activities out and contribute to the PAG.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over, receiving care for Long Covid symptoms at one of the participating LC sites.
* Willing and able to consent for their data to be used for research and/or service evaluation purposes. Consent will be gathered via patient information sheet and formal recording of consent (on the phone application).

Exclusion Criteria:

* Inability to independently complete electronic or paper-based outcome measures, questionnaires or other research-based paperwork.
* Unable to give Informed Consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred into one of the ten Long Covid services by their General Practitioner (GP), or other clinicians (Positive Antigen or Antibody test is not required.)
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
European Quality of Life Five Dimensions | 2 years
  Quality of Life VAS score min 0 max 100
COVID-19 Yorkshire Rehabilitation Scale | 2 years
  Symptom severity (min 0 max 100) and functional disability (min 0 max 50) and health state (min 0 max 10)

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Sivan, MD, Principal Investigator — University of Leeds
Locations (1):
- University of Leeds, Leeds, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Horton M, Smith AB, Milne R, Winch D, Rayner C, Halpin S, O'Connor R, Rocha Lawrence R, Greenwood DC, Bakerly ND, Evans R, Kwon J, Dawes H, Wood C, Williams P, Master H, Mansoubi M, De Kock JH, Mullard J, Ormerod M, Mir G, Petrou S, O'Connor DB, Sivan M; LOCOMOTION Consortium. Large-Scale Psychometric Assessment and Validation of the Modified COVID-19 Yorkshire Rehabilitation Scale Patient-Reported Outcome Measure for Long COVID or Post-COVID Syndrome. J Med Virol. 2026 Feb;98(2):e70816. doi: 10.1002/jmv.70816. PMID 41586458
- [Derived] Lee C, Williams P, Abrahams A, Darbyshire J, Davies HE, De Kock J, Esmer U, Jones SA, Newey V, Scott J, Smith N, Winch D, Master H, Elkin S; LOCOMOTION Consortium. What Can We Learn Four Years On? A Multi-Centre Service Evaluation Exploring Symptoms, Functional Impact, Recovery and Care Pathways in Long Covid. Health Expect. 2025 Dec;28(6):e70435. doi: 10.1111/hex.70435. PMID 41199609
- [Derived] Mullard J, Mir G, Herbert C, Evans S; LOCOMOTION Consortium. 'You're just a Guinea pig': Exploring the barriers and impacts of living with long COVID-19: A view from the undiagnosed. Sociol Health Illn. 2024 Nov;46(8):1602-1625. doi: 10.1111/1467-9566.13795. Epub 2024 Jun 8. PMID 38850204
- [Derived] Greenhalgh T, Darbyshire JL, Lee C, Ladds E, Ceolta-Smith J. What is quality in long covid care? Lessons from a national quality improvement collaborative and multi-site ethnography. BMC Med. 2024 Apr 15;22(1):159. doi: 10.1186/s12916-024-03371-6. PMID 38616276
- [Derived] Lee C, Greenwood DC, Master H, Balasundaram K, Williams P, Scott JT, Wood C, Cooper R, Darbyshire JL, Gonzalez AE, Davies HE, Osborne T, Corrado J, Iftekhar N, Rogers N, Delaney B, Greenhalgh T, Sivan M; LOCOMOTION Consortium. Prevalence of orthostatic intolerance in long covid clinic patients and healthy volunteers: A multicenter study. J Med Virol. 2024 Mar;96(3):e29486. doi: 10.1002/jmv.29486. PMID 38456315
- [Derived] Mullard JCR, Kawalek J, Parkin A, Rayner C, Mir G, Sivan M, Greenhalgh T. Towards evidence-based and inclusive models of peer support for long covid: A hermeneutic systematic review. Soc Sci Med. 2023 Mar;320:115669. doi: 10.1016/j.socscimed.2023.115669. Epub 2023 Jan 14. PMID 36708608
- [Derived] Sivan M, Greenhalgh T, Darbyshire JL, Mir G, O'Connor RJ, Dawes H, Greenwood D, O'Connor D, Horton M, Petrou S, de Lusignan S, Curcin V, Mayer E, Casson A, Milne R, Rayner C, Smith N, Parkin A, Preston N, Delaney B; LOCOMOTION consortium. LOng COvid Multidisciplinary consortium Optimising Treatments and servIces acrOss the NHS (LOCOMOTION): protocol for a mixed-methods study in the UK. BMJ Open. 2022 May 17;12(5):e063505. doi: 10.1136/bmjopen-2022-063505. PMID 35580970